CLINICAL TRIAL: NCT03600532
Title: Testing the Efficacy of the Teachable Moment Brief Intervention for Suicide Attempt Survivors in an Inpatient Setting: Effects on Psychosocial and Experimental Pain Outcomes
Brief Title: Teachable Moment Brief Intervention for Suicide Attempt Survivors in an Inpatient Setting
Acronym: TMBI-IP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to lack of participant recruitment
Sponsor: University of Tulsa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TU1808
Record Dates: First submitted 2018-07-03; First posted 2018-07-26 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Suicide, Attempted
Keywords: experimental pain
MeSH Terms: conditions — Suicide, Attempted

STUDY DESIGN:
Intervention Model Description: Participants will be assigned in even numbers to TMBI & TAU or recruited as part of a CCG
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Teachable Moment Brief Intervention (Experimental): The TMBI is informed by evidence based strategies to collaboratively identify 1) drivers of suicidal ideation, 2) functional aspects of the recent suicide attempt, 3) the patient's relationship with the concept of suicide, 4) what has been lost and gained as a result of the suicide attempt, 5) short term management suicide prevention management strategies, and 6) documentation of factors to address in a suicide-specific treatment plan.
  Interventions: Behavioral: Teachable Moment Brief Intervention (TMBI)
- Treatment as Usual (TAU) (No Intervention): Usual care at Laureate Psychiatric Clinic and Hospital Adult Stabilization Unit who have attempted suicide involves psychiatric evaluation/treatment and ongoing medical stabilization. Patients will engage in usual care or a rest period before completing the post-assessment.
- Community Control Group (CCG) (No Intervention): Patients will engage in a rest period before completing the post-assessment.

INTERVENTIONS:
Behavioral: Teachable Moment Brief Intervention (TMBI) — Behavioral intervention informed by Collaborative Assessment and Management of Suicidality and Dialectical Behavior Therapy/Cognitive Behavior Therapy to assist in positive recovery trajectory following a suicide attempt.
  Arms: Teachable Moment Brief Intervention

SUMMARY:
This study is looking at the helpfulness of a brief treatment targeting suicidality (Teachable Moment Brief Intervention [TMBI]) and experimental pain responses in an inpatient population as well as collecting comparison data from the community.

DETAILED DESCRIPTION:
The proposed study will use an innovative one-session psychotherapeutic intervention called the Teachable Moment Brief Intervention (TMBI) for suicide attempters admitted to a psychiatric inpatient unit. A total of 60 patients will be recruited from the inpatient psychiatry unit at Laureate Psychiatric Clinic and Hospital and 30 healthy community members for the study. Informed consent will be obtained for all participants and administration of the baseline assessment battery will be completed prior to randomization for patients. Patients will then be randomized to either (a) an experimental group receiving TMBI or (b) a group receiving treatment as usual (TAU). The intervention will consist of no more than 90 minutes (expected mean is 45 minutes for the intervention based upon previous studies of the TMBI) of 1:1 interaction with a study clinician. All participants will complete a follow-up assessment immediately following TMBI, TAU, or a rest period. Further, patients receiving the experimental intervention will then be asked to complete a client satisfaction survey. The aim will be to assess whether TMBI affects psychological, experimental pain, and autonomic nervous system responses as compared to TAU and community controls.

ELIGIBILITY:
TMBI & TAU (data collection at Laureate Psychiatric Clinic and Hospital [LPCH])

Inclusion:

-admitted to LPCH subsequent to a suicide attempt

Exclusion:

* acute psychosis,
* inability to read English, or
* taking narcotic or opioid pain medication

CCG (data collection in the Psychophysiology Laboratory for Affective Neuroscience [PLAN] on the University of Tulsa campus)

Exclusion:

* acute psychosis,
* current suicide ideation,
* history of self-harm,
* inability to read English, or
* taking narcotic or opioid pain medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Changes in Beck Scale for Suicide Ideation | Assessed immediately before the intervention or rest period (baseline) and immediately after the intervention or rest period (approximately 1 hour from baseline)
  19-item assessment used to evaluate the current intensity of the patient's specific attitudes toward, behavior, and plans to commit suicide. Total score will be reported which ranges from 0 (no suicidal ideation) to 38 (high suicidal ideation).

SECONDARY OUTCOMES:
Changes in Stages of Change Questionnaire | Assessed immediately before the intervention or rest period (baseline) and immediately after the intervention or rest period (approximately 1 hour from baseline)
  18-item measure that measures motivation to engage in treatment/work on problems. Total score will be summed from all items, with range from 18 (low motivation) to 90 (high motivation). Four subscales will also be reported as follows: Precontemplation ranges from 5 (low) to 25 (high) with higher scores indicating higher motivation. Contemplation ranges from 4 (low) to 20 (high) with higher scores indicating higher motivation. Action ranges from 5 (low) to 25 (high) with higher scores indicating higher motivation. Maintenance ranges from 4 (low) to 20 (high) with higher scores indicating higher motivation.
Changes in Reasons for Living Inventory | Assessed immediately before the intervention or rest period (baseline) and immediately after the intervention or rest period (approximately 1 hour from baseline)
  48-item measure that rates the importance of different reasons why people choose not to kill themselves. Total score will be reported, which ranges from 48 (low reasons for living) to 288 (High reasons for living).
Changes in Adult State Hope Scale | Assessed immediately before the intervention or rest period (baseline) and immediately after the intervention or rest period (approximately 1 hour from baseline)
  6-item measure of ongoing self-directed thinking. Total score will be reported, which ranges from 6 (low hope) to 48 (high hope).
Change in Positive and Negative Affect Schedule | Assessed immediately before the intervention or rest period (baseline) and immediately after the intervention or rest period (approximately 1 hour from baseline)
  20-item self-report measure of Positive (PANAS-PA; 10 items) and Negative (PANAS-NA; 10 items) Affect. Each PANAS emotion word is rated on a 5-point scale, 1 (very slightly) to 5 (extremely) corresponding to the extent to which each emotion is experienced at the time of administration. Thus, higher scores indicate more and/or stronger positive (PANAS-PA) or negative (PANAS-NA) emotions.
Changes in Ischemic Pain Outcomes | Assessed immediately before the intervention or rest period (baseline) and immediately after the intervention or rest period (approximately 1 hour from baseline)
  Ischemia produces a pain akin to clinical musculoskeletal pain syndromes. 120 handgrip exercises will be conducted at a rate of 1/sec at 50% maximal effort using a dynamometer (handgrip force meter), and then the arm will be raised to promote exsanguination. A blood pressure cuff will then be inflated around the arm biceps to 220 mm/Hg to produce ischemia. The participants will be instructed to inform the experimenter when they first experience pain (pain threshold). The cuff will be deflated when the pain is no longer tolerable or after 3 minutes (pain tolerance). After 3 minutes as measured by a stopwatch (or when the participant discontinues the task), they will be asked to rate the average and peak pain intensity during the task on a scale from 0 (no pain) to 100 (intolerable pain).
Changes in Mechanical Pressure Pain Outcomes | Assessed immediately before the intervention or rest period (baseline) and immediately after the intervention or rest period (approximately 1 hour from baseline)
  Delivered using von Frey hairs (i.e., monofilament = brush with only one bristle) on the back of the nondominant hand. The monofilament, sized 6.45, will be applied to the skin at a 90 degree angle, which exerts 180 grams of force. The participant will be asked to rate their pain on a scale of 0 (no pain) to 100 (intolerable pain).
Changes in Temporal Summation of Pain | Assessed immediately before the intervention or rest period (baseline) and immediately after the intervention or rest period (approximately 1 hour from baseline)
  Delivered using von Frey hairs (i.e., monofilament = brush with only one bristle) on the back of the nondominant hand. The 6.45 monofilament will be applied to the skin at a 90 degree angle 10 times, once per second. The participant will be asked to rate their peak pain during these 10 stimuli on a scale of 0 (no pain) to 100 (intolerable pain). Temporal summation is the extent by which pain experience increases over the course of repeated stimulus presentation. Therefore, it will be measured as the difference between the peak pain over the course of these 10 stimuli and the rating of the single stimulus (mechanical pressure pain).
Changes in Skin Conductance Level | Assessed immediately before the intervention or rest period (baseline) and immediately after the intervention or rest period (approximately 1 hour from baseline)
  Sympathetic arousal will be measured from skin conductance level (SCL), measured from a BioDerm meter (UFI Model 2701) and corresponding electrodes filled with isotonic paste and placed on the volar surface of the medial digit on the index and middle fingers of the left hand. SCL will be assessed during the resting BP measurement prior to any testing, for one minute prior to pain testing during the BP measurement, during pain testing, and for one minute following pain testing during the second BP measurement. SCL will be recorded every 15 seconds manually by the experimenter. A pain-related change score will be created to find the difference between the average SCL during baseline and during pain testing. A recovery-related change score will be created to find the difference between average SCL during pain testing and the average post pain testing SCL.
Changes in Blood Pressure | Assessed immediately before the intervention or rest period (baseline) and immediately after the intervention or rest period (approximately 1 hour from baseline)
  Resting systolic and diastolic blood pressure (BP) will be measured using a medical blood pressure monitor prior to testing. BP will also be measured just prior to and immediately following the pain testing. BP will be measured on the right arm. A pain-related change score will be created to find the difference between the BP before and after pain testing.
Changes in Cardiovascular Measurements | Assessed immediately before the intervention or rest period (baseline) and immediately after the intervention or rest period (approximately 1 hour from baseline)
  Resting heart rate (HR; e.g., beats per minute [BPM]) will be measured using a medical blood pressure monitor prior to testing. HR will also be measured just prior to and immediately following the pain testing. HR will be measured on the right arm. A pain-related change score will be created to find the difference between the HR before and after pain testing.

CONTACTS AND LOCATIONS:
Overall Officials: Cassandra A Sturycz, MA, Principal Investigator — University of Tulsa
Locations (2):
- United States (2):
  - University of Tulsa, Psychophysiology Laboratory for Affective Neuroscience (PLAN), Tulsa, Oklahoma
  - Laureate Psychiatric Clinic and Hospital, Tulsa, Oklahoma

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617